CLINICAL TRIAL: NCT03044119
Title: A Comparative Evaluation of the Effect of Platelet Rich Fibrin Matrix With and Without Peripheral Blood Mesenchymal Stem Cells on Implant Stability : A Randomized Controlled Clinical Trial
Brief Title: The Effect of Platelet Rich Fibrin Matrix With and Without Peripheral Blood Mesenchymal Stem Cells on Implant Stability
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: KLE Society's Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr Laveena Singhal, Dr Laveena, KLE Society's Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KLESInstitute
Record Dates: First submitted 2017-02-02; First posted 2017-02-06 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Dental Implants
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Intervention Model Description: The selected sites would be randomly (coin toss method) assigned into an edentulous area allowing for the placement of a minimum of two adjacent dental implants being randomly assigned into (G1) - Dental implant with PRFM and (G2) - Dental implant with peripheral blood mesenchymal stem cells embedded in PRFM.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The selected sites would be randomly (coin toss method) assigned into an edentulous area .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dental Implant with PRFM (Active Comparator): Intervention in the form of Dental Implants placement in the adjacent edentulous bone with the placement of platelet rich fibrin matrix a biological material procured from patient's peripheral blood
  Interventions: Biological: Dental Implant with PRFM
- Dental Implant with PRFM and PBMSCs (Experimental): Intervention in the form of Dental Implant placement in the adjacent edentulous bone with the placement of platelet rich fibrin matrix and peripheral blood mesenchymal stem cells which are the biological materials procured from patient's peripheral blood
  Interventions: Biological: Dental Implant with PRFM and PBMSCs

INTERVENTIONS:
Biological: Dental Implant with PRFM — placement of a minimum of two adjacent dental implants being randomly assigned into (G1) - Dental implant with PRFM
  Arms: Dental Implant with PRFM
Biological: Dental Implant with PRFM and PBMSCs — placement of a minimum of two adjacent dental implants being randomly assigned into (G2) - Dental implant with peripheral blood mesenchymal stem cells embedded in PRFM.
  Arms: Dental Implant with PRFM and PBMSCs

SUMMARY:
The Primary Objectives of the present study are :

* To Evaluate the effect of platelet rich fibrin matrix (PRFM) and peripheral blood mesenchymal stem cells (PBMSCs) on implant stability.
* To Compare the effect of platelet rich fibrin matrix (PRFM) alone to peripheral blood mesenchymal stem cells (PBMSCs) embedded in platelet rich fibrin matrix (PRFM) on implant stability.

DETAILED DESCRIPTION:
The addition of molecules or growth factors to the implant surface is an approach to enhance bone to implant contact (BIC).1 Platelet rich fibrin matrix (PRFM) is an autologous concentrated platelet-rich thrombin free fibrin matrix, prepared by two step centrifugation of blood. Platelets isolated, remain intact and retain their growth factor compliment. This allows a more effective, sustained release of growth factors to the wound site following PRFM application.2 During the second spin, a cross-linking of fibrin takes place, resulting in the formation of a dense fibrin matrix, within which a concentration of viable platelets can be found. Having an organized fibrin matrix at the start of healing accelerates the speed of vascular ingress into the wound compared to non-accelerated healing, which requires a longer time for fibrin formation and the development of vascularity. The earlier the vascularity is established, faster is the migration of the bone-forming cells at the wound site and initiation of bone formation. Therapeutic applications of platelet-rich products have led to improved bone regeneration and faster titanium implant osseointegration, which improve the stability and maintenance of dental implants by increasing BIC.1 Mesenchymal stem cells (MSCs) is a multipotent stromal cell with prominent regenerative functions. MSCs were first identified and isolated from bone marrow and then found in various tissues including umbilical cord, adipose tissue and peripheral blood. Among these sources peripheral blood MSCs draw increasing attention as they share similar biological characteristics with MSCs derived from bone marrow or adipose tissue. Bone marrow derived mesenchymal stem cells(BMMSCs) are multipotent cells capable of differentiating into osteoblasts, chondrocytes, adipocytes , fibroblasts, tenocytes, and myoblasts , which are considered as a cell source for various tissue repair and regenerating bone defects.3 The requirements of aspiration of bone marrow from the patient will cause pain and morbidity of the donor sites. It will be very convenient if peripheral blood mesenchymal stem cells (PBMSCs) could be harvested and expanded to enough numbers, with their osteogenic capacity maintained in a clinical permitted period.

The literature search does not show any human clinical trial conducted till date to assess the regenerative potential of this new modality i.e. PRFM and peripheral blood mesenchymal stem cells. This study therefore aims at the evaluation of PRFM and PBMSCs as regenerative materials for implant stability.

ELIGIBILITY:
Inclusion Criteria:

* Patient with age group between 25-50 years
* Radiographic imaging(IOPA/OPG/CBCT/RVG) of the area of interest showing sufficient residual bone volume to receive two or more adjacent implants of ≥ 3.5 mm in diameter and 11.0 mm in length
* Extraction at least 6 months prior to the study.

Exclusion Criteria:

* Para-functional habits
* Smoking more than 10 cigarettes per day
* Excessive consumption of alcohol
* Patient's with systemic diseases contraindicated for surgery
* Localized radiotherapy, Antitumor chemotherapy of the oral cavity
* Liver, blood, and/or kidney diseases
* Immunosuppression
* Current corticosteroid or bisphosphonate use;
* Pregnancy
* Mucocutaneous diseases involving the oral cavity and
* Poor oral hygiene.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-07-20 (Estimated); Study Completion 2019-10-20 (Estimated)

PRIMARY OUTCOMES:
Insertion torque values at the time of placement of dental implant | on the implant placement day
  insertion torque values will be recorded during the day of placement of implants.

SECONDARY OUTCOMES:
Implant stability quotient (ISQ) using Resonance frequency analysis (RFA). | 3 months
  Implant stability quotient (ISQ) using Resonance frequency analysis (RFA) with the help of Osstell device at 1 week, 1 month and 3 months post operatively

CONTACTS AND LOCATIONS:
Overall Officials: Sudhir R Patil, MDS, Principal Investigator — KLE Society's Institute of Dental Sciences
Locations (1):
- Kle Society'S Institute of Dental Sciences, Bengaluru, Karnataka, India

IPD SHARING:
Plan to Share IPD: Yes
in the form of research publication